CLINICAL TRIAL: NCT03086083
Title: Bilateral Brain Stimulation in Trauma Therapy: a Randomized Clinical Trial
Brief Title: Bilateral Brain Stimulation in Trauma Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ciclo de Mutação (Other)
Collaborators: Sao Jose do Rio Preto Medical School (Other)
Responsible Party: Principal Investigator, Maria Aparecida Junqueira Zampieri, Clinical Supervisor, Principal Investigator, Ciclo de Mutação
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 0000-0002-5442-4488
Record Dates: First submitted 2017-02-18; First posted 2017-03-22 (Actual); Last update posted 2017-03-28 (Actual); Status verified 2017-03

CONDITIONS: Intervention Study; Handling (Psychology)
Keywords: Traumatic memories; comparative study; single session; EMDR; Beck inventory
MeSH Terms: interventions — Clinical Protocols

STUDY DESIGN:
Intervention Model Description: A randomized, parallel, before-after, blind study was performed. Thirty nine subjects were randomly distributed to two groups: one session of EMDR psychotherapy standard and other with EMDR standard protocol without its typical brain bilateral stimulation. The results of the Beck scales for anxiety, depression and hopelessness and the impact of events test were compared between groups.
Who Masked: Participant, Outcomes Assessor
Masking Description: All participants was invited to one session of brief Psychotherapy with a new model.
  To the outcome assessor was said to study if was significant difference between those data from two groups α e β.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EMDR standard protocol (Experimental): Standard EMDR protocol, once.
  Interventions: Behavioral: EMDR standard protocol
- protocol without brain stimulation (Active Comparator): Standard EMDR protocol without brain stimulation, once
  Interventions: Behavioral: protocol without brain stimulation

INTERVENTIONS:
Behavioral: EMDR standard protocol — Patient have only one standard EMDR session about a traumatic situation remembered by him.
  Arms: EMDR standard protocol
Behavioral: protocol without brain stimulation — Patient have only one standard EMDR session about a traumatic situation remembered by him, however, without the bilateral brain stimulation.
  Other Names: EMDR altered protocol
  Arms: protocol without brain stimulation

SUMMARY:
Comparatively studied the effects of Eye Movement Desensitization and Reprocessing (EMDR) bilateral brain stimulation in trauma therapy.

A randomized, parallel, before-after, blind study was performed.

DETAILED DESCRIPTION:
Comparatively studied the effects of Eye Movement Desensitization and Reprocessing (EMDR) bilateral brain stimulation in trauma therapy.

A randomized, parallel, before-after, blind study was performed. Thirty nine subjects were randomly distributed to two groups: one session of EMDR psychotherapy standard and other with EMDR standard protocol without its typical brain bilateral stimulation. The results of the Beck scales for anxiety, depression and hopelessness and the impact of events test were compared between groups.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria for the study were to be a university student, over 18 years old, to have a complaint associated to a traumatic life event and to have accepted to participate of the study.

Exclusion Criteria:

* Exclusion criteria were the existence of untreated psychiatric disorders and the hypothesis of worsening of the subject's status as the number of sessions in this study was restricted to once.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-10-21 (Actual); Primary Completion 2015-03-13 (Actual); Study Completion 2015-08-28 (Actual)

PRIMARY OUTCOMES:
Impact of Events Test | Before and immediately after the psychotherapy session, which has average of 1:30 hours.
  Self-administered questionnaire to measure Impact of the traumatic event, which the patient have selected for this intervention
Beck scale for anxiety | Before and immediately after the psychotherapy session, which has average of 1:30 hours.
  Self-administered questionnaire to measure anxiety, in this case, when the patient are thinking about that specific traumatic event, which he or she selected for this intervention.

SECONDARY OUTCOMES:
Change from baseline Beck scale for depression at the final of session | Before and immediately after the conclusion of the session, which has average of 1:30 hours
  Self-administered questionnaire to measure depression, in this case, when the patient are thinking about that specific traumatic event, which he or she select for this intervention.
Change from baseline Beck scale for hopelessness at the final of session | Before and immediately after the conclusion of the session, which has average of 1:30 hours
  Self-administered questionnaire to measure hopelessness

CONTACTS AND LOCATIONS:
Overall Officials: Maria Aparecida J Zampieri, Ph.D., Principal Investigator — Ciclo de Mutação; Marina J Zampieri, Graduate, Study Chair — Ciclo de Mutação; Alexandre J Zampieri, Graduate, Study Chair — Ciclo de Mutação; Moacir F Godoy, Ph.D., Study Chair — Sao Jose do Rio Preto Medical School
Locations (1):
- Ciclo de Mutação: Psychotherapy and Research, São José do Rio Preto, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Nazari H, Momeni N, Jariani M, Tarrahi MJ. Comparison of eye movement desensitization and reprocessing with citalopram in treatment of obsessive-compulsive disorder. Int J Psychiatry Clin Pract. 2011 Nov;15(4):270-4. doi: 10.3109/13651501.2011.590210. Epub 2011 Aug 3. PMID 22122001
- [Result] Shapiro F, Maxfield L. Eye Movement Desensitization and Reprocessing (EMDR): information processing in the treatment of trauma. J Clin Psychol. 2002 Aug;58(8):933-46. doi: 10.1002/jclp.10068. PMID 12115716
- [Result] Shapiro F. The role of eye movement desensitization and reprocessing (EMDR) therapy in medicine: addressing the psychological and physical symptoms stemming from adverse life experiences. Perm J. 2014 Winter;18(1):71-7. doi: 10.7812/TPP/13-098. PMID 24626074
- [Result] Ronconi JM, Shiner B, Watts BV. Inclusion and exclusion criteria in randomized controlled trials of psychotherapy for PTSD. J Psychiatr Pract. 2014 Jan;20(1):25-37. doi: 10.1097/01.pra.0000442936.23457.5b. PMID 24419308
- [Result] Herkt D, Tumani V, Gron G, Kammer T, Hofmann A, Abler B. Facilitating access to emotions: neural signature of EMDR stimulation. PLoS One. 2014 Aug 28;9(8):e106350. doi: 10.1371/journal.pone.0106350. eCollection 2014. PMID 25165974
- [Result] Rimini D, Molinari F, Liboni W, Balbo M, Daro R, Viotti E, Fernandez I. Effect of Ocular Movements during Eye Movement Desensitization and Reprocessing (EMDR) Therapy: A Near-Infrared Spectroscopy Study. PLoS One. 2016 Oct 26;11(10):e0164379. doi: 10.1371/journal.pone.0164379. eCollection 2016. PMID 27783688
- See also: Universidade Estadual Paulista Julio de Mesquita Filho - UNESP STAEPE - Seção Tecnica de Apoio ao Ensino, Pesquisa e Extensão Instituto de Biociências, Letras e Ciências Exatas / IBILCE / UNESP — http://www.fapesp.br/
- See also: The EMDR International Association (EMDRIA) is a professional association where EMDR practitioners and EMDR researchers seek the highest standards for the clinical use of EMDR therapy. — http://www.emdria.org/
- See also: The EMDR Brazilian Association is a association where EMDR practitioners and EMDR researchers seek standards for the clinical use of EMDR therapy. — http://www.emdr.org.br/